CLINICAL TRIAL: NCT05895266
Title: A Phase 1 Open-Label Drug-Drug Interaction Study Between ABBV-903 and Midazolam
Brief Title: A Study to Assess Drug-Drug Interaction Between ABBV-903 and Midazolam in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-225
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-903; Midazolam
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: Period 1 (Experimental): In Period 1 on Day 1, participants will receive liquid midazolam.
  Interventions: Drug: Midazolam
- Part 1: Period 2 (Experimental): In Period 2 on Day 1, participants will receive ABBV-903 oral tablets. In Period 2 on Day 10, participants will receive liquid midazolam and ABBV-903 oral tablets. Participants will be followed-up for approximately 30 days.
  Interventions: Drug: ABBV-903; Drug: Midazolam
- Part 2: Period 1 (Experimental): In Period 1 on Day 1, participants will receive liquid midazolam.
  Interventions: Drug: Midazolam
- Part 2: Period 2 (Experimental): In Period 2 on Day 1, participants will receive ABBV-903 oral tablets. In Period 2 on Day 5, participants will receive liquid midazolam and ABBV-903 oral tablets. Participants will be followed-up for approximately 30 days.
  Interventions: Drug: ABBV-903; Drug: Midazolam

INTERVENTIONS:
Drug: ABBV-903 — Oral Tablet
  Arms: Part 1: Period 2; Part 2: Period 2
Drug: Midazolam — Oral Liquid

SUMMARY:
The main objective of this study is to assess the drug-drug interaction and pharmacokinetics of ABBV-903 and Midazolam in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI is ≥ 18.0 to ≤ 32 kg/m2 after rounding to the tenth.
* Negative test result for SARS-CoV-2 infection upon initial confinement
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), endocrine, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of diseases aggravated or triggered by ultraviolet radiation and no history of abnormal reaction photosensitivity or photoallergy to sunlight, or artificial source of intense light, especially ultraviolet light.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 40 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum Plasma Concentration (Cmax) of ABBV-903 | Up to approximately 40 days
  Cmax of ABBV-903
Maximum Plasma Concentration (Cmax) of Midazolam | Up to approximately 40 days
  Cmax of midazolam
Maximum Plasma Concentration (Cmax) of 1-OH-Midazolam | Up to approximately 40 days
  Cmax of 1-OH-midazolam
Time to Cmax (Tmax) of ABBV-903 | Up to approximately 40 days
  Tmax of ABBV-903
Time to Cmax (Tmax) of Midazolam | Up to approximately 40 days
  Tmax of midazolam
Time to Cmax (Tmax) of 1-OH-Midazolam | Up to approximately 40 days
  Tmax of 1-OH-midazolam
Terminal Phase Elimination Half-Life (t1/2) of ABBV-903 | Up to approximately 40 days
  Terminal phase elimination half-life of ABBV-903
Terminal Phase Elimination Half-Life (t1/2) of Midazolam | Up to approximately 40 days
  Terminal phase elimination half-life of midazolam
Terminal Phase Elimination Half-Life (t1/2) of 1-OH-Midazolam | Up to approximately 40 days
  Terminal phase elimination half-life of 1-OH-midazolam
Area Under the Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUCt) of ABBV-903 | Up to approximately 40 days
  AUCt of ABBV-903
Area Under the Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUCt) of Midazolam | Up to approximately 40 days
  AUCt of midazolam
Area Under the Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUCt) of 1-OH-Midazolam | Up to approximately 40 days
  AUCt of 1-OH-midazolam
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-903 | Up to approximately 40 days
  AUCinf of ABBV-903
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of Midazolam | Up to approximately 40 days
  AUCinf of midazolam
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of 1-OH-Midazolam | Up to approximately 40 days
  AUCinf of 1-OH-midazolam

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 254970, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-225